CLINICAL TRIAL: NCT06860737
Title: A Randomized Clinical Trial on the Effectiveness of Novel Spectacle Lenses for Myopia Prevention in Pre-myopic Children
Brief Title: A Randomized Clinical Trial on the Effectiveness of Novel Plano Spectacle Lenses on Myopia Prevention in Pre-myopic Children
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Eye Disease Prevention and Treatment Center (Other)
Collaborators: Essilor International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: WS10405
Record Dates: First submitted 2025-03-02; First posted 2025-03-06 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-03

CONDITIONS: Myopic Children
Keywords: pre-myopic children; evaluation; intervention; comliance

STUDY DESIGN:
Intervention Model Description: Children aged 6-9 years old with pre-myopia are randomly assigned to a control group and an intervention group at a 1:1 ratio. The intervention group uses novel plano spectacle lenses for at least 8 hours a day, and the control group doesn't receive any intervention. The efficacy of novel plano spectacle lenses in delaying myopia onset in pre-myopia children is evaluated by comparing the one-year incidence of myopia onset between intervention group and control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Use of novel plano spectacle lenses for at least 8 hours a day with objective wearing time measured by smart frame and objective outdoor time measured by smart bracelet.
  Interventions: Device: Novel plano spectacle lenses
- Control group (No Intervention): Objectively measuring outdoor time by smart bracelet.

INTERVENTIONS:
Device: Novel plano spectacle lenses — Use of novel plano spectacle lenses for at least 8 hours a day with objective wearing time measured by smart frame and objective outdoor time measured by smart bracelet.
  Arms: Intervention group

SUMMARY:
Evaluate the efficacy, safety and wearing time compliance of novel plano spectacle lenses in delaying myopia onset in pre-myopic children and provide scientific basis for the development of myopia prevention strategies for children.

DETAILED DESCRIPTION:
Children aged 6-9 years old with pre-myopia are randomly assigned to a control group and an intervention group at a 1:1 ratio. The intervention group uses novel plano spectacle lenses for at least 8 hours a day, and the control group doesn't receive any intervention. The efficacy of novel plano spectacle lenses in delaying myopia onset in pre-myopia children is evaluated by comparing the one-year incidence of myopia onset between intervention group and control group.

ELIGIBILITY:
Inclusion Criteria:

* At the time of signing the informed consent form, the subject's age must be ≥6 years and <10 years (6-9.99 years);
* Both eyes are not myopic (SE>-0.50D under cycloplegia) and at least one eye meets the pre-myopia condition ( -0.50D< SE under cycloplegia ≤+0.75D); [spherical equivalent (SE)=Sph+Cyl/2]
* Astigmatism ≤1.00D in each eye;
* Difference in SER (Anisometropia) between the two eyes should not exceed ≤1.50D;
* Unaided distance and near visual acuity of at least 0.1 logMAR in each eye ;
* Be in good general health;
* Be able to actively cooperate with the intervention plan and ophthalmological examination;
* Normal binocular vision
* At least one parent with SER ≤-3.00 D

Exclusion Criteria:

* Incapable of expressing consent
* All categories of persons particularly protected by law
* Subject in another study which might have an influence on vision or interfere with study assessment.
* Previous use of other prevention solutions, such as but not limited to red light therapy within 6 months, Atropine and other interventions were used within 3 months;
* History or presence of an ocular disease, systemic disease, strabismus or amblyopia or other binocular vision abnormalities, accommodation dysfunction, cataract and eye surgery;
* Those who are allergic cycloplegic drugs;
* Other reasons that the investigator considers inappropriate for inclusion in the study.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 388 (Estimated)
Dates: Start 2025-03-15 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
One-year cumulative myopia incidence in either eye | From enrollment to the end of intervention for one year
  One-year cumulative myopia incidence in either eye

SECONDARY OUTCOMES:
Changes of spherical equivalent under cycloplegia | From enrollment to the end of intervention for one year
  Changes of spherical equivalent under cycloplegia
Changes of axial length | From enrollment to the end of intervention for one year
  Changes of axial length
Changes of choroidal thickness | From enrollment to the end of intervention for one year
  Changes of choroidal thickness
Changes of unaided distance visual acuity | From enrollment to the end of intervention for one year
  Changes of unaided distance visual acuity
Changes of visual acuity with novel spectacle lenses and Single Vision spectacle lenses | From enrollment to the end of intervention for one year
  Changes of visual acuity with novel spectacle lenses and Single Vision spectacle lenses
Changes of accommodation function | From enrollment to the end of intervention for one year
  Changes of accommodation function
Wearing time recorded in the questionnaire and smart frame | From enrollment to the end of intervention for one year
  Wearing time recorded in the questionnaire and smart frame
Objective outdoor time recorded with smart bracelet | From enrollment to the end of intervention for one year
  Objective outdoor time recorded with smart bracelet

OTHER OUTCOMES:
Incidence and severity of adverse events (AEs) related to study intervention | From enrollment to the end of intervention for one year
  Incidence and severity of adverse events (AEs) related to study intervention
Monocular best-corrected visual acuity (BCVA) | From enrollment to the end of intervention for one year
  Monocular best-corrected visual acuity (BCVA)
Assessment of symptoms, complaints related to the study intervention, as reported by participants. | From enrollment to the end of intervention for one year
  Assessment of symptoms, complaints related to the study intervention, as reported by participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangui He, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang J, Du L, Chen J, Zhang B, Yang J, Du Y, Gao W, Zou H, Xu X, He X. A randomized clinical trial on the effectiveness of plano spectacle lenses with lenslets on myopia prevention in pre-myopic children: Study protocol of a randomized controlled trial. Acta Ophthalmol. 2025 Sep 21. doi: 10.1111/aos.70007. Online ahead of print. PMID 40976937